CLINICAL TRIAL: NCT03410134
Title: Clinical Evaluation of Vital Pulp Therapy in Young Permanent Molars With Irreversible Pulpitis
Brief Title: Assessment of Vital Pulp Therapy in Permanent Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Irreversible pulpitis
Record Dates: First submitted 2017-12-03; First posted 2018-01-25 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries Extending to Pulp; Pulp Disease, Dental
Keywords: Permanent teeth; Vital pulp therapy; MTA
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoMTA (Experimental): Vital pulp therapy with NeoMTA
  Interventions: Device: NeoMTA

INTERVENTIONS:
Device: NeoMTA — NeoMTA™ Plus® root and pulp treatment material is a powder/gel system with no resin. The components are an extremely fine powder primarily tricalcium and dicalcium silicate plus a water-based gel.

SUMMARY:
The purpose of this study is to evaluate the long term clinical performance of vital pulp therapy of young permanent teeth with irreversible pulpitis

DETAILED DESCRIPTION:
Permanent molar teeth meeting the inclusion criteria will be included into the study. Following local anaesthesia and dental dam application, caries excavation will be performed; and after exposure, the pulp will be amputated to the level of the canal orifices (full pulpotomy) using a sterile high-speed round bur under water coolant. After haemostasis is achieved, Mineral trioxide aggregate (MTA) will be gently placed over the pulp to a thickness of 2-3 mm and the tooth will be restored using glass ionomer cement and composite resin. A postoperative periapical radiograph will be taken. Patients will be reviewed at 6., 12., 24. and 36. months for clinical and radiographical success. The data will be analysed statistically using chi square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of the patients who accept to participate and sign the informed consent
* Patients who have at least one vital permanent molar teeth with irreversible pulpitis symptoms
* Teeth which can be restorable after the treatment.
* Teeth which has good periodontal health and in the absence of sinus tracts or swelling.

Exclusion Criteria:

* Patients and parents of the patients who does not accept to participate and sign the informed consent
* Teeth which have dentoalveolar or extraoral swelling
* Teeth which have periodontal disease, mobility or alveolar bone loss
* Teeth which are not restorable
* Patients who are not cooperative with the treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation of vital pulp therapy in permanent teeth with irreversible pulpitis | 3 years
  Long-term success of vital pulp therapy in young permanent teeth with irreversible pulpitis. Evaluation criteria will be;
  1. spontaneous pain (absent/present);
  2. tenderness to percussion/palpation (absent/present);
  3. mobility (no mobility/ 1mm/ 2mm/ 3mm mobility)
  4. swelling (absent/present);
  5. fistula (absent/present)
  6. periapical/interradicular radiolucency (absent/present);
  7. widened periodontal ligament (absent/present);
  8. loss of lamina dura (absent/present);
  9. internal/external root resorption (absent/present).

CONTACTS AND LOCATIONS:
Overall Officials: Zafer C Cehreli, DDS,PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asgary S, Eghbal MJ, Ghoddusi J, Yazdani S. One-year results of vital pulp therapy in permanent molars with irreversible pulpitis: an ongoing multicenter, randomized, non-inferiority clinical trial. Clin Oral Investig. 2013 Mar;17(2):431-9. doi: 10.1007/s00784-012-0712-6. Epub 2012 Mar 21. PMID 22431145
- [Background] Taha NA, Ahmad MB, Ghanim A. Assessment of Mineral Trioxide Aggregate pulpotomy in mature permanent teeth with carious exposures. Int Endod J. 2017 Feb;50(2):117-125. doi: 10.1111/iej.12605. Epub 2016 Jan 30. PMID 26715408
- [Background] Qudeimat MA, Alyahya A, Hasan AA. Mineral trioxide aggregate pulpotomy for permanent molars with clinical signs indicative of irreversible pulpitis: a preliminary study. Int Endod J. 2017 Feb;50(2):126-134. doi: 10.1111/iej.12614. Epub 2016 Feb 22. PMID 26841969